CLINICAL TRIAL: NCT07202598
Title: A Phase 2 Randomized Stepped Wedge Study of Emapalumab in APECED Enteritis
Brief Title: Randomized Stepped Wedge Study of Emapalumab in APECED Enteritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002480; 002480-I
Record Dates: First submitted 2025-10-01; First posted 2025-10-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12-08

CONDITIONS: Autoimmune Polyendocrinopathy Candidiasis Ectodermal Dystrophy Enteritis
Keywords: Autoimmune Polyendocrinopathy Candidiasis Ectodermal Dystrophy
MeSH Terms: conditions — Polyendocrinopathies, Autoimmune | interventions — Emapalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): No observation period prior to start of study drug.
  Interventions: Drug: Emapalumab
- Group 2 (Experimental): 2 month observation period prior to start of study drug.
  Interventions: Drug: Emapalumab
- Group 3 (Experimental): 4 month observation period prior to start of study drug.
  Interventions: Drug: Emapalumab
- Group 4 (Experimental): 6 month observation period prior to start of study drug.
  Interventions: Drug: Emapalumab

INTERVENTIONS:
Drug: Emapalumab — Emapalumab will be administered via IV infusion once a month. The initial dose of emapalumab is 3 mg/kg followed by a second dose of 3 mg/kg after 3 days. Subsequently, the dose is 3 mg/kg once a month for five additional doses.

SUMMARY:
Background:

Autoimmune polyendocrinopathy-candidiasis-ectodermal dystrophy (APECED), also known as Autoimmune polyendocrine syndrome type-1 (APS-1), is a disease that causes the immune system to attack parts of a person s body. In some people, APECED attacks the small intestine; this causes an illness called enteritis.

Objective:

To test a drug (emapalumab) in people with enteritis caused by APECED.

Eligibility:

People aged 2 to 75 years with APECED and enteritis. They must also be enrolled in protocol 11-I-0187.

Design:

Participants will have 10-13 study visits in an 18-month period.

Participants will be screened. They will have a physical exam with blood tests. These tests will be repeated at every study visit. They will have a test of their heart function. This will be at screening and prior to drug administration.

Other tests are optional: Participants may have imaging exams and a test of lung function. They may have an endoscopy, which is an exam of their digestive tract. Participants may provide samples of urine, stool, nail clippings, saliva, vaginal fluid, or skin. Photos may be taken of their skin or scalp. These tests may be repeated at some visits.

Emapalumab is given through a tube attached to a needle inserted into a vein. All participants will receive 7 doses: 2 on their first study visit; then 1 each at 30-day intervals. Some participants will have an observation period before they begin taking the drug; in those situations, they will either be seen in person or via video visit every 2 months before starting emapalumab to see how their symptoms change over time.

Participants will have a follow-up visit 1 month after their last dose. Then they will have 2 telehealth visits at 30-day intervals. They will have a final clinic visit 1 year after their first dose.

...

DETAILED DESCRIPTION:
Study Description:

This is a phase 2 randomized stepped wedge open-label study to evaluate the efficacy and safety of the anti-interferon-gamma (IFN-gamma) monoclonal antibody, emapalumab, in autoimmune polyendocrinopathycandidiasis-ectodermal dystrophy (APECED) enteritis. Qualifying participants will be randomized to initiate emapalumab at 0, 2, 4, or 6 months post-baseline visit. They will be admitted for up to 10 days for an inpatient visit to start receiving emapalumab in 2 intravenous (IV) infusions 3 days apart. Thereafter, participants will receive 5 additional monthly IV infusions of emapalumab followed by an additional in-person visit 1 month after the final dose of emapalumab. All participants will be followed for an additional 6 months after this via virtual visits every 2 months and an in-person visit at the end of this 6-month period. Throughout the study, participants will be monitored for adverse events (AEs) and will complete patient-reported outcome (PRO) metrics to track their symptoms and general wellbeing as well as have blood draws for safety labs and research.

Primary Objective:

To evaluate the efficacy of emapalumab on gastrointestinal (GI) symptoms as measured by the APECED enteritis score (APECED ES) in participants with APECED enteritis.

Secondary Objectives:

1. To evaluate the safety of emapalumab in participants with APECED enteritis.
2. To assess additional measures of efficacy related to amelioration of intestinal dysfunction in response to emapalumab treatment.
3. To investigate the effect of emapalumab on PROs related to GI symptoms.
4. To evaluate the effect of emapalumab on histologic and immunologic features of the GI tract.

Exploratory Objectives:

1. To investigate the effect of emapalumab on improving clinical symptoms and associated laboratory, histologic, and immunologic abnormalities in affected organs and tissues beyond the GI tract.
2. To investigate the effect of emapalumab on PROs of affected organs and tissues beyond the GI tract.
3. To investigate the effect of emapalumab on prevention of development of new APECED-associated complications during the treatment period.
4. To examine the effects of emapalumab on ameliorating immunologic readouts of excessive IFN-gamma/JAK/STAT signaling in peripheral blood and affected organs and tissues beyond the GI tract.
5. To determine whether emapalumab treatment affects the composition of microbial communities at the mucocutaneous barriers.
6. To describe the pharmacokinetics (PK) of emapalumab in this population.

Primary Endpoint:

Averaged changes in APECED ES from baseline.

Secondary Endpoints:

1. Incidence of serious adverse events (SAEs), AEs requiring study drug discontinuation, and other AEs during the 6 months of emapalumab treatment.
2. Change from baseline in APECED ES at 6 months after emapalumab initiation.
3. Averaged changes in irritable bowel syndrome (IBS) QOL score from baseline.
4. Change from baseline in IBS QOL score at 6 months after emapalumab initiation.
5. Averaged changes in scores for 36-Item Short Form Health Survey (SF-36) for adult participants or Pediatric Quality of Life Inventory (PedsQL) for pediatric participants from baseline.
6. Changes from baseline in SF-36 (adults) or PedsQL (pediatrics) at 6 months after emapalumab initiation.
7. Averaged changes in serum zinc from baseline in participants with decreased zinc at baseline.
8. Changes from baseline in serum zinc at 6 months after emapalumab initiation in participants with decreased zinc at baseline.
9. Change from baseline in 48-hour fecal fat at 6 months after emapalumab initiation in participants with elevated fecal fat at baseline.
10. Change from baseline in histologic and immunologic abnormalities of duodenal tissue after 6 months of treatment.
11. Averaged changes in serum CXCL9 from baseline.
12. Change from baseline in serum CXCL9 at 6 months after emapalumab initiation.

Exploratory Endpoints:

1. Incidence of SAEs, AEs requiring study drug discontinuation, and other AEs during the 6 months after emapalumab treatment ends.
2. Change from baseline in APECED ES at 2 months after emapalumab initiation.
3. Change from baseline in APECED ES at 4 months after emapalumab initiation.
4. Time from emapalumab initiation that participants achieved a mean 50% reduction in APECED ES.
5. Proportion of participants achieving a 50% reduction in APECED ES at 2, 4, and 6 months after emapalumab initiation.
6. Proportion of participants with a 50% increase in APECED ES at 2, 4, and 6 months after completion of 6 months of emapalumab treatment (change is based on measurement at completion of 6 months of treatment).
7. Averaged changes in fecal calprotectin from baseline in participants with elevated calprotectin at baseline.
8. Change from baseline in fecal calprotectin at 6 months after emapalumab initiation in participants with elevated calprotectin at baseline.
9. Change from baseline in fraction of unconjugated bile acids out of total bile in 48-hour stool collection at 6 months after emapalumab initiation in participants with elevated unconjugated bile acids >10% of total fecal bile acids at baseline.
10. Averaged changes in serum zinc from baseline in all participants.
11. Changes from baseline in serum zinc at 6 months after emapalumab initiation in all participants.
12. Time to development of next APECED-associated manifestation during the 6 months of emapalumab treatment.
13. Number of APECED-associated manifestations that developed during the 6 months of emapalumab treatment.
14. Change from baseline in histologic or immunologic abnormalities of oral, esophageal, and gastric mucosal tissues at 6 months after emapalumab initiation.
15. Change from baseline in histologic or immunologic abnormalities of salivary gland tissue in participants with Sjogren's-like syndrome at 6 months after emapalumab initiation.
16. Change from baseline in salivary flow rate in participants with Sjogren's-like syndrome at 6 months after emapalumab initiation.
17. Change from baseline in histologic or immunologic abnormalities of scalp tissue in participants with alopecia at 6 months after emapalumab initiation.
18. Change from baseline in Severity of Alopecia Tool (SALT) score in participants with alopecia areata at 6 months after emapalumab initiation.
19. Change in clinician-reported outcome (ClinRO) measures for eyelash and eyebrow presence from baseline at 6 months after emapalumab initiation.
20. Change from baseline in nail appearance in participants with nail dystrophy at 6 months after emapalumab initiation.
21. Change in ClinRO and PRO measures for nail appearance from baseline at 6 months after emapalumab initiation.
22. Change from baseline in Vitiligo Area Scoring Index (VASI) in participants with vitiligo at 6 months after emapalumab initiation.
23. Change from baseline in the oral, vaginal, stool, and/or skin microbiome at 6 months after emapalumab initiation.
24. Change from the 6-month pre-treatment baseline in the number of urticarial episodes in participants with urticaria during the 6 months of emapalumab treatment.
25. Change from baseline in corticosteroid dose requirements, adrenocorticotropic hormone, cortisol, electrolyte, and renin levels in participants with adrenal insufficiency at 6 months after emapalumab initiation.
26. Change from baseline in calcium replacement requirements, intact parathyroid hormone, and calcium levels in participants with hypoparathyroidism at 6 months after emapalumab initiation.
27. Change from baseline in thyroid hormone replacement dose requirements, thyroid-stimulating hormone, free and total thyroxine, anti-thyroglobulin, and thyroid peroxidase antibody in participants with hypothyroidism at 6 months after emapalumab initiation.
28. Change from baseline in insulin requirements, hemoglobin A1C, fasting glucose, insulin, C-peptide, urine ketone, and glucose levels in participants with type-1 diabetes at 6 months after emapalumab initiation.
29. Change from baseline in levels of follicle-stimulating hormone, estradiol, anti-Mullerian hormone, total and free testosterone, and sex hormone-binding globulin in participants with hypogonadism at 6 months after emapalumab initiation.
30. Change from baseline in Ocular Surface Disease Index (OSDI) in participants with dry eyes at 6 months after emapalumab initiation.
31. Change from baseline measure corneal fluorescein staining (grading scale), tear breakup time (TBUT) (seconds), automated keratography TBUT, and tear meniscus assessments in participants with keratoconjunctivitis at 6 months after emapalumab initiation.
32. Change from baseline grade of conjunctival redness in participants with keratoconjunctivitis at 6 months after emapalumab initiation.
33. Change from baseline in tear production as assessed by Schirmer's test in participants with Sjogren's-like syndrome at 6 months after emapalumab initiation.
34. Change from the 6-month pre-treatment baseline in the number of oral and/or vaginal candidiasis infections during the 6 months of emapalumab treatment.
35. Change in clinical and radiographic manifestations of joint abnormalities in participants with arthritis at 6 months after emapalumab initiation.
36. Change in respiratory symptoms, radiographic abnormalities, and pulmonary function test (PFT) and 6-minute walk (6MW) parameters in participants with pneumonitis at 6 months after emapalumab initiation.
37. Change in liver function test in participants with hepatitis at 6 months after emapalumab initiation.
38. Change in renal function test in participants with tubulointerstitial nephritis at 6 months after emapalumab initiation.
39. Change in fecal pancreatic elastase-1 and serum fat-soluble vitamins in participants with exocrine pancreatic insufficiency at 6 months after emapalumab initiation.
40. Change from the 6-month pre-treatment baseline in the number of chronic inflammatory demyelinating polyneuropathy flares in affected participants during the 6 months of emapalumab treatment.
41. Change from baseline in titers of cytokine- and tissue-specific autoantibodies at 6 months after emapalumab initiation.
42. Change from baseline of levels of phosphorylated STAT molecules in peripheral blood mononuclear cells (PBMCs) at 6 months after emapalumab initiation.
43. Change from baseline in serum CXCL9 at 2 months after emapalumab initiation.
44. Change from baseline in serum CXCL9 at 4 months after emapalumab initiation.
45. Averaged changes in serum CXCL10 from baseline.
46. Change from baseline in serum CXCL10 at 2 months after emapalumab initiation.
47. Change from baseline in serum CXCL10 at 4 months after emapalumab initiation.
48. Change from baseline in serum CXCL10 at 6 months after emapalumab initiation.
49. Change from baseline in transcriptional profile in whole blood and tissue biopsies at 6 months after emapalumab initiation.
50. Measurements of serum concentration of emapalumab to evaluate the PK of the study drug in participants with APECED.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participant must be able to understand and provide informed consent.
  2. Aged >= 2 to <= 75 years.
  3. Currently co-enrolled on NIH protocol 11-I-0187, "The Natural History and Pathogenesis of Human Fungal Infections."
  4. Patients with APECED (genetic or clinical diagnosis) and enteritis (with APECED ES > 50 at screening).
  5. Duration of enteritis greater than 6 months.
  6. Is naive or unresponsive to other treatments for enteritis.
  7. Willingness to use acyclovir or valacyclovir prophylaxis for the prevention of herpes viral reactivation.
  8. Willingness to use entecavir prophylaxis against hepatitis B virus reactivation, if applicable.
  9. Vaccinations should be up to date in agreement with current Centers for Disease Control and Prevention immunization guidelines prior to start of emapalumab.
  10. Proficient in written English.
  11. Participants who can get pregnant or impregnate their partner must agree to use at least one highly effective method of contraception when engaging in sexual activities that can result in pregnancy, starting at screening until 12 weeks after the last dose. Highly effective contraceptive measures include:
* Stable use of combined (estrogen- and progestogen-containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) starting 1 month prior to screening.
* Intrauterine device (IUD); intrauterine hormone-releasing system.
* Two barrier methods (e.g., condom with spermicide, diaphragm with spermicide, or cervical cap and spermicide). Internal and external condoms may not be used together.
* Bilateral tubal ligation.

Periodic abstinence (calendar, symptothermal, and post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception.

EXCLUSION CRITERIA:

1. Known history of hypersensitivity to emapalumab.
2. History of active intestinal disease other than enteritis such as inflammatory bowel disease.
3. Current or recent use of any investigational drug (within 3 months or 5 half-lives, whichever is longer, prior to screening).
4. Scheduled to participate in another clinical study involving an investigational drug during the course of this study.
5. History of alcohol or drug abuse within 6 months prior to screening.
6. Presence of one or more of the following clinically significant laboratory abnormalities:

   1. Serum ALT >= 3 times upper limit of normal (ULN).
   2. Serum total bilirubin >= 2 times ULN.
   3. Serum creatinine >= 2 times ULN.
7. Planned or anticipated major surgical procedure during the study.
8. Plans to receive any live or live attenuated vaccines within 1 month of the anticipated first dose of emapalumab.
9. Known or suspected immunodeficiency disorder besides APECED.
10. History of untreated invasive opportunistic infections (e.g., tuberculosis, non-tuberculous mycobacterial infections, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystis pneumonia, aspergillosis) despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged infections suggesting an immune-compromised status as judged by the investigator.
11. Untreated latent tuberculosis infection.
12. Infection with HIV.
13. Untreated infection with hepatitis B or C.
14. History of serious bacterial infection within the last 3 months prior to screening, unless treated and resolved with antibiotics, or any chronic bacterial infection (e.g., chronic pyelonephritis, osteomyelitis).
15. Current pregnancy or breastfeeding.
16. Past or current medical problems or findings from physical examination, EKG, or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Averaged changes in APECED ES from baseline. | Duration of study
  To evaluate the efficacy of emapalumab on gastrointestinal (GI) symptoms as measured by the APECED enteritis score (APECED ES) in participants with APECED enteritis.

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs), AEs requiring study drug discontinuation, and other AEs during the 6 months of emapalumab treatment. | Duration of study
  To evaluate the safety of emapalumab in participants with APECED enteritis.
Change from baseline in APECED ES at 6 months after emapalumab initiation. | Duration of study
  To assess additional measures of efficacy related to amelioration of intestinal dysfunction in response to emapalumab treatment.
Averaged changes in irritable bowel syndrome (IBS) QOL score from baseline and change from baseline in IBS QOL score at 6 months after emapalumab initiation. | Duration of study
  To investigate the effect of emapalumab on PROs related to GI symptoms.
Averaged changes in scores for 36-Item Short Form Health Survey (SF-36) for adult participants or Pediatric Quality of Life Inventory (PedsQL) for pediatric participants from baseline and changes from baseline in SF-36 (adults) or PedsQL (pediat... | Duration of study
  To investigate the effect of emapalumab on PROs related to GI symptoms.
Averaged changes in serum zinc from baseline in participants with decreased zinc at baseline and changes from baseline in serum zinc at 6 months after emapalumab initiation in participants with decreased zinc at baseline. | Duration of study
  To evaluate the effect of emapalumab on histologic and immunologic features of the GI tract.
Change from baseline in 48-hour fecal fat at 6 months after emapalumab initiation in participants with elevated fecal fat at baseline. | Duration of study
  To evaluate the effect of emapalumab on histologic and immunologic features of the GI tract.
Change from baseline in histologic and immunologic abnormalities of duodenal tissue after 6 months of treatment. | Duration of study
  To evaluate the effect of emapalumab on histologic and immunologic features of the GI tract.
Averaged changes in serum CXCL9 from baseline and change from baseline in serum CXCL9 at 6 months after emapalumab initiation. | Duration of study
  To evaluate the effect of emapalumab on histologic and immunologic features of the GI tract.

CONTACTS AND LOCATIONS:
Overall Officials: Michail S Lionakis, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared in open-access or restricted-access data repositories, as appropriate for the type of data.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002480-I.html